CLINICAL TRIAL: NCT01824329
Title: Prospective Phase II Randomized Trial of Prostate Capsule Sparing Cystectomy and Nerve-sparing Radical Cystoprostatectomy in Men With Bladder Cancer
Brief Title: Prostate Capsule Sparing Cystectomy and Nerve-sparing Radical Cystoprostatectomy in Men With Bladder Cancer
Acronym: SPARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alon Weizer, Associate Professor, Urology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00000769
Record Dates: First submitted 2013-03-31; First posted 2013-04-04 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Bladder Cancer; Transitional Cell Carcinoma of the Bladder
Keywords: Bladder Cancer; Transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostate capsule sparing cystectomy Group (Active Comparator): Prostate capsule sparing cystectomy involves removing the entire bladder.
  Interventions: Procedure: Prostate capsule sparing cystectomy
- Nerve sparing cystectomy Group (Active Comparator): Nerve sparing cystectomy involves removal of the whole bladder and the entire prostate.
  Interventions: Procedure: Nerve sparing cystectomy

INTERVENTIONS:
Procedure: Prostate capsule sparing cystectomy — Removes the adenoma and prostatic urethra along with the urinary bladder, but leaves in situ the prostatic capsule and subsequently the surrounding neurovascular bundle.
  Arms: Prostate capsule sparing cystectomy Group
Procedure: Nerve sparing cystectomy — Attempts to spare the cavernosal nerves that travel immediately adjacent to the lateral prostate and are routinely divided during a standard RCP.
  Arms: Nerve sparing cystectomy Group

SUMMARY:
Bladder cancer is the 4th most common cancer amongst men. If bladder cancer invades the muscle of the bladder or fails local treatments, surgical removal of the bladder (cystectomy) with creation of a new bladder from intestine is required. However, standard cystectomy affects urinary function and sexual function. The investigators are evaluating two modifications to cystectomy to determine to what extent they preserve urinary and sexual function.

DETAILED DESCRIPTION:
Radical cystoprostatectomy (RCP) is the standard treatment of muscle invasive, and refractory high grade, superficial bladder cancer. RCP involves the removal of the bladder and prostate. While this is an effective treatment for patients with organ confined disease almost all men following RCP are impotent due to resection of the neurovascular bundles that control erectile dysfunction. While neobladders (new bladders formed out of detubularized bowel connected to the native urethra) allow patients to void normally, many of these patients have difficulty with urinary incontinence. Two modifications have been developed to improve the functional outcomes of this surgery. Nerve sparing cystectomy (NSC) attempts to spare the cavernosal nerves that travel immediately adjacent to the lateral prostate and are routinely divided during a standard RCP. Published series of NSC have shown improved preservation of sexual function and less urinary incontinence without compromising cancer control. Another alternative, prostate capsule sparing cystectomy (PCSC), removes the adenoma and prostatic urethra along with the urinary bladder, but leaves in situ the prostatic capsule and subsequently the surrounding neurovascular bundle. Several retrospective series have demonstrated preservation of sexual function and improved urinary continence compared to standard RCP and neobladder. A concern with PCSC is that prostate or urothelial cancer invading the prostate could be left behind with preservation of the prostate capsule. Most reported series in which patients were screened with digital rectal exam, prostate and prostatic urethral biopsy, and PSA blood testing could identify patients at risk for having prostate or urothelial cancer in the prostate capsule preoperatively to recommend an alternative approach. Therefore, both NSC and PCSC appear to offer better urinary and sexual function in properly selected patients over conventional RCP in retrospective series. However, these procedures have not been evaluated prospectively in a randomized fashion. Our intent is to evaluate the functional outcomes of PCSC and NSC with orthotopic neobladder in terms of urinary and sexual function using the bladder cancer index, a validated quality of life instrument, and determine the surgical margin status, and complications of the two surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be men 18 years or older
* histologic diagnosis of Ta - T2 transitional cell carcinoma within 3 months of enrollment.
* no nodal or metastatic disease on pre-operative CT or MRI within 3 months of enrollment.
* no evidence of malignancy in the prostate based on 12-core transrectal ultrasound guided prostate needle biopsy and transurethral resection of prostatic urethra16
* candidate for and willingness to undergo a radical cystectomy and orthotopic neobladder by the urologic surgeon performing the procedure.
* competent to provide informed consent
* able to read and write English
* willing to be randomized to PCSC versus NSC.

Exclusion Criteria:

* histologically proven stage T3 or greater bladder cancer and/or evidence of metastatic disease by work-up described above.
* creatinine > 2.2 mg/dl.
* refuse to complete study requirements.
* prior pelvic radiation to bladder or prostate.
* history of radical prostatectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Post-operative urinary function | 7 years
  Assess post-operative urinary function using the bladder cancer index (BCI) in patients randomized to either prostate capsule sparing cystectomy (PCSC) or nerve sparing radical cystoprostatectomy (NSC).

SECONDARY OUTCOMES:
Bladder cancer control | 7 years
  Determine bladder cancer control with PCSC compared to NSC as measured by margin status and time to disease recurrence.
Sexual function | 7 Years
  Determine sexual function after PCSC and NSC using the BCI.
Adverse event rates | 7 years
  Determine adverse event rates after PCSC and NSC.
Peri-operative differences | 7 years
  Determine peri-operative differences between PCSC and NSC in terms of operative time, estimated blood loss, length of hospital stay, and time to catheter removal.

CONTACTS AND LOCATIONS:
Overall Officials: Alon Weizer, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States